CLINICAL TRIAL: NCT05206084
Title: A Prospective, Multi-Center, Single-Blinded, Randomized Trial of the Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System in Patients With Coronary Artery Disease: IRONMAN-II
Brief Title: A Clinical Investigation to Evaluate the Safety and Efficacy of IBS in Patients With Coronary Artery Disease
Acronym: IRONMAN-II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotyx Medical (Shenzhen) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IBS II
Record Dates: First submitted 2021-12-20; First posted 2022-01-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBS (Experimental): Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System
  Interventions: Device: Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System (IBS)
- XIENCE (Active Comparator): Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System
  Interventions: Device: Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System (IBS) — Subjects in this arm will be treated with IBS
  Arms: IBS
Device: Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System — Subjects in this arm will be treated with XIENCE
  Arms: XIENCE

SUMMARY:
A prospective, multi-center, single-blinded, randomized trial to assess the safety and efficacy of the Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System (IBS) in treating patients with coronary artery disease compared to the Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System (XIENCE).

DETAILED DESCRIPTION:
IRONMAN-II is a prospective, multi-center, single-blinded, randomized trial to assess the safety and efficacy of the Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System (IBS) in treating patients with coronary artery disease compared to the Abbott Vascular XIENCE Everolimus Eluting Coronary Stent System (XIENCE). A total of 518 subjects with coronary artery lesion(s) are intended to participate in this study. Angiographic follow-up will be required at 2 years, and an OCT subset including 50 subjects will undergo OCT follow-up. Clinical follow-up will be required at postoperative, 1 month, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years. The primary endpoint is late lumen loss at 2 years.

The primary objective of this trial is to support the China pre-market approval of IBS Sirolimus-Eluting Iron Bioresorbable Coronary Scaffold System. IRONMAN-II will evaluate the safety and efficacy of the IBS in treating patients with coronary artery disease. The primary endpoint is late lumen loss at 2 years.

The powered secondary objective is to evaluate long-term vascular function and patency of the IBS treated segments compared to XIENCE treated segments. The powered secondary endpoints include Quantitative Flow Ratio (QFR) and cross-section level mean flow area measured by OCT for OCT subset at 2 years.

Data from the primary endpoint and two powered secondary endpoints will evaluate the non-inferiority of the IBS as compared to XIENCE.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must between 18 and 75 years old, male or non-pregnant female.
2. Patient must have evidence of myocardial ischemia (e.g., stable, unstable angina, silent myocardial ischemia, or acute myocardial infarction>1 week) suitable for elective PCI.
3. One or two de novo target lesions each located in a different epicardial vessel.

   1. If there is one target lesion, another non-target lesion may be treated but the non-target lesion must be present in a different epicardial vessel, and must be treated first with a successful result prior to randomization of the target lesion.
   2. If two target lesions are present, they must be present in different epicardial vessels and both satisfy the angiographic eligibility criteria.
   3. The definition of epicardial vessels means the left anterior descending artery (LAD), the left circumflex artery (LCX), and the right coronary artery (RCA) and their branches. Thus, for example, the subject must not have lesions requiring treatment in both the LAD and a diagonal branch.
4. Lesion(s) must have a visually estimated length of ≤33mm, diameter between range of 2.5-4.0mm, and each lesion can be completely covered by a stent.
5. Lesion(s) must have a visually estimated diameter stenosis of ≥70% (or ≥50% and have evidence of myocardial ischemia in this location) with a TIMI flow of ≥1.
6. Patient can understand the study purpose, voluntarily participate in the study, sign the informed consent, and willing to undergo protocol-required invasive angiographic follow-ups.

Exclusion Criteria:

* General Exclusion Criteria

  1. Patient had an acute myocardial infarction (AMI) or CK and CK-MB have not returned to within normal limits after myocardial infarction within 7 days of the index procedure.
  2. Patient has implanted stent in the target vessel within 1 year of the index procedure, or is scheduled to undergo re-intervention in the future 6 months.
  3. Patient with a history of coronary artery bypass (coronary artery bypass grafting).
  4. Patient with contraindications on coronary artery bypass graft surgery.
  5. Patient with severe heart failure (NYHA class ≥III) or left ventricular ejection fraction<40% (by echocardiography or contrast left ventriculography).
  6. Patient with known renal insufficiency: serum creatinine > 2.0 mg/dl or 177 μmol/L, or/and patient on dialysis.
  7. Patient with known hepatic insufficiency: ALT, AST >3 times the upper limit of normal.
  8. Patient had an ischemic stroke within 6 months or transient ischemic neurological attack (TIA) within 3 months before the index procedure, or has tendency of hypercoagulation as per investigator judgement or laboratory test.
  9. Patient with bleeding diathesis, active gastrointestinal ulcers, history of cerebral hemorrhage or subarachnoid hemorrhage, contraindications on antiplatelet agents and anticoagulant therapy, and unable to undergoing antithrombotic therapy.
  10. Patient with known allergy to aspirin, clopidogrel, heparin, contrast agent, PDLLA, sirolimus and metal (iron, zinc etc).
  11. Patient with a history of disease related to iron overload or iron disorder, such as hereditary hemochromatosis, etc.
  12. Patient with life expectancy <2 years.
  13. Patient is already participating in another drug or medical device clinical trial that has not yet reached its primary endpoint.
  14. Patient with poor compliance and cannot comply with the protocol requirement as per investigator judgement.
  15. Subject has received a heart transplant.
  16. Patient with unstable arrhythmia, such as high-risk ventricular premature beat and ventricular tachycardia.
  17. Patient requires chemotherapy for malignancy.
  18. Patient with known immunosuppressive or autoimmune disease, and is receiving or scheduled to receive immunosuppressant therapy.
  19. Patient is receiving or scheduled to receive chronic anticoagulation therapy such as aspirin and warfarin, etc.
  20. Patient is scheduled to receive a surgery that requires to stop antiplatelet drugs such as heparin and clopidogrel within 6 months after the index procedure.
  21. Patient has a platelet count <100x10^9/L or >700 x10^9/L, a white blood cell count of <3 x10^9/L during the screening period.
  22. Patient with diffuse peripheral vascular disease, and cannot use 6F catheter.
  23. Patient with prior valvular surgery.
* Angiographic exclusion criteria

  1. Chronic total occlusion (TIMI flow of 0 before the index procedure).
  2. Target lesion is located in left main.
  3. Aorto-ostial lesion (within 3 mm of the ostium).
  4. Target lesion involving a bifurcation lesion with side branch ≥2.5 mm in diameter (the ostium of side branch has restenosis ≥40% or require balloon pre-dilatation).
  5. Visible thrombus in target vessels.
  6. Severe triple vessels lesions and all require revascularization.
  7. Severe calcified or distorted lesions which unable to predilate, not suitable for stent delivery and expansion, impair delivery including:

     1. Extreme angulation (≥ 90°) proximal to or within the target lesion
     2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion
     3. Moderate or heavy calcification proximal to or within the target lesion
  8. In-stent restenosis target lesion.
  9. Target lesion involves a myocardial bridge.
  10. The investigational stent would need to cross the previously implanted stent to reach the target lesion.
  11. Target lesion which prevents complete balloon pre-dilatation, defined as full balloon expansion with the following outcomes:

      1. Residual diameter stenosis (DS%) is < 40% (per visual estimation), ≤ 20% is strongly recommended.
      2. TIMI flow of 3 (per visual estimation).
      3. No angiographic complications (e.g., distal embolization, side branch closure).
      4. No dissections National Heart, Lung, and Blood Institute (NHLBI) grade D-F.
      5. No chest pain lasting > 5 minutes.
      6. No ST depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
In-segment Late lumen loss (LLL) | 2 years

SECONDARY OUTCOMES:
Powered Secondary Endpoint: Quantitative Flow Ratio (QFR) | 2 years
Powered Secondary Endpoint: Cross-section level mean flow area measured by OCT | 2 years
  Only for subjects in OCT subset
Rate of Device Success | Immediately post-procedure
  Device Success is defined as: A visually estimated diameter stenosis of < 30% after implantation of the device and TIMI flow of III.
Rate of Lesion Success | Immediately post-procedure
  Lesion Success is defined as: The attainment of visual residual stenosis < 30% and TIMI flow of III after any intervention in target lesion.
Rate of Clinical Success | ≤ 7 days post the index procedure (In-hospital )
  Clinical Success is defined as: lesion success, AND there is no major adverse cardiac event in the hospitalization period.
Rate of Device-oriented Composite Endpoint (DoCE) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
  Target Lesion Failure (TLF), defined as the composited endpoints of cardiac death/Target Vessel Myocardial Infarction (TV-MI)/Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Rate of Patient-oriented Composite Endpoint (PoCE) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
  Including all-cause mortality, any myocardial infarction and any revascularization.
Rate of Death (Cardiac, Vascular and Non-cardiovascular) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
Rate of Myocardial infarction (Attributable to target vessel (TV-MI),or Not attributable to target vessel (NTV-MI)) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
Rate of Target Lesion Revascularization (Ischemia driven, or not ischemia driven) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
Rate of Target Vessel Revascularization (Ischemia driven, or not ischemia driven) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
Rate of all coronary revascularization | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
Rate of Stent Thrombosis defined by ARC (definite and probable) | 1 Month, 6 Months, 1 Year, 2 Years, 3 Years, 4 Years, 5 Years
  Stent thrombosis is defined by Academic Research Consortium (ARC) criteria as definite, probable, and possible. Stent thrombosis was categorized as acute, Subacute, late, very late.
Acute recoil | Immediately post-procedure
Minimal lumen diameter (MLD) (In-stent, in-segment, proximal 5mm and distal 5mm MLD) | at post-procedure, 2 years
Diameter stenosis (DS %) (In-device, in-segment, proximal 5mm and distal 5mm DS%) | at post-procedure, 2 years
Late Lumen Loss (LLL) (In-device, proximal 5mm and distal 5mm LLL) | 2 years
Angiographic binary restenosis (ABR) (In-device, in-segment, proximal 5mm and distal 5mm ABR) | 2 years
Thickness of neointima (struts level) | 2 years
Minimal lumen area | 2 years
Percentage of neointima-covered struts | 2 years
Late incomplete strut apposition | 2 years
Lumen area stenosis % | 2 years
Healing score | 2 years
  Healing score = (presence of intra-scaffold structure * 4) + (presence of both malapposed and uncovered struts * 3) + (presence of uncovered struts alone * 2) + (presence of malapposition alone * 1).
Stent Absorption (%) | 2 years
Late recoil area | 2 years
Late recoil proportion | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Yunnan Cardiovascular Hospital, Kunming, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gao R, Song L, Fu G, Guan C, Li Y, Jia S, He Y, Chen J, Qi F, Yu M, Yang B, Zhang Y, Zhang Z, He S, Chen Y, Ma Y, Zhou Y, Wang L, Zhao G, Qian J, Guo N, Sun Z, Huang Y, Li W, Wang Y, Ge J, Han Y, Stone GW; IRONMAN II Investigators. Sirolimus-Eluting Iron Bioresorbable Scaffolds vs Everolimus-Eluting Stents for Percutaneous Coronary Intervention: A Randomized Trial (IRONMAN II). J Am Coll Cardiol. 2026 Feb 11:S0735-1097(25)10492-0. doi: 10.1016/j.jacc.2025.12.024. Online ahead of print. PMID 41670556